CLINICAL TRIAL: NCT02111239
Title: Preoperative Imagining in DIEP Flap Breast Reconstruction: A Randomized Controlled Trial Evaluating Cost and Patient-Reported Outcomes
Brief Title: Preoperative Imaging in DIEP Flap Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sunnybrook106-2011
Record Dates: First submitted 2013-08-01; First posted 2014-04-11 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: DIEP; DIEP flap; Breast reconstruction; Breast Cancer; CTA; MRA
MeSH Terms: conditions — Breast Neoplasms | interventions — Computed Tomography Angiography; Magnetic Resonance Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No imaging (No Intervention): No preoperative imaging is performed for this group
- CTA (Experimental): Patients randomized to this group will undergo a preoperative CTA scan.
  Interventions: Device: CTA
- MRA (Experimental): Patients randomized to this group will undergo a preoperative MRA scan.
  Interventions: Device: MRA

INTERVENTIONS:
Device: CTA — pelvic/abdominal CTA scan
  Other Names: preoperative CTA; computed tomography angiography
  Arms: CTA
Device: MRA — pelvic/abdominal MRA scan
  Other Names: preoperative MRA; magnetic resonance angiogram
  Arms: MRA

SUMMARY:
The purpose of this study is to determine whether preoperative abdominal imaging using either CT angiogram (CTA), or MR angiogram (MRA) will impact perforator dissection time, cost, and patient outcomes in DIEP flap breast reconstruction.

DETAILED DESCRIPTION:
This study will prospectively compare the clinical, economic and patient outcomes of preoperative imaging using either CTA or MRA with those of no preoperative imaging in patients undergoing deep inferior epigastric perforator (DIEP) flap breast reconstruction. Subjects will randomly undergo either a CTA scan or an MRA scan, or no scan (control) preoperatively. An operative plan based on perforator size and course will be devised by an interventional radiologist and a plastic surgeon. The DIEP flap procedure will be planned for controls.

Subjects will not be told if the operative plan is changed intraoperatively. Flap dissection time and changes in operative plan will be recorded intraoperatively and surgeon stress will be evaluated following surgery. Pain and narcotic use will be evaluated preoperatively and on days 1-4 postoperatively. The Breast-Q will be completed preoperatively and at 3 weeks, 3 months and 12 months postoperatively. Groups will be compared in terms of all variables measured.

ELIGIBILITY:
Inclusion Criteria:

* candidate for DIEP flap breast reconstruction
* speak/read/write English
* have undergone or will undergo unilateral or bilateral mastectomy

Exclusion Criteria:

* previous abdominal surgery that may preclude a DIEP flap reconstruction
* active smoker
* BMI over 35
* severe claustrophobia
* sensitivity to intravenous CT contrast medium (Visipaque 320) or MR contrast medium (Gadovist 1.0)
* urgency of surgery that precludes study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Time for flap dissection | 1 day - during surgery
  Time to reach exposure of perforators combined with time for flap elevation will be recorded during the surgical procedure.
Change in BREAST-Q Scores | Preoperatively, Postoperatively at 3 weeks, 3 months, 12 months
  Self-administered quality of life and outcomes questionnaire for women that undergo breast reconstruction.

SECONDARY OUTCOMES:
Whether change in operative procedure occurred during surgery | 1 day
  Change of operative plan either prior to surgery as a result of preoperative imaging, or intra-operatively, will be recorded
Change in Memorial Pain Assessment Card (MPAC) Scores | Baseline, postoperatively on the first 4 days, and at 3 weeks, 3 months and 12 months
  Self-administered questionnaire consisting of 4 questions related to pain, pain relief, and mood.
NASA-Task Load Index (TLX) | once - immediately postoperatively
  Completed by the operating surgeon to evaluate workload based on 6 scales: mental demand, physical demand, temporal demand, performance, effort and frustration.
Economic Outcome | 1 year
  The costs of medical imaging and operating expenses will be calculated and compared between study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Lipa, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada